CLINICAL TRIAL: NCT05182645
Title: MBMCrohn: Die Wirkung Eines Stressreduktion- Und Lebensstilmodifikations-programms Auf Die Lebensqualität Von Patienten Mit Morbus Crohn- Eine Machbarkeitsstudie
Brief Title: Effect of a Stress Reduction and Lifestyle Modification Programme on the Quality of Life of Crohn's Disease Patients
Acronym: MBMCrohn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jost Langhorst (Other)
Collaborators: Sozialstiftung Bamberg (Other); University of Wuerzburg (Other); Wuerzburg University Hospital (Other); Bavarian State Ministry of Health and Care (Other Government)
Responsible Party: Sponsor-Investigator, Jost Langhorst, Clinical Professor, Universität Duisburg-Essen
Organization: Universität Duisburg-Essen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19096
Record Dates: First submitted 2020-08-11; First posted 2022-01-10 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: Waiting Control Group Design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lifestyle-modification (Experimental): Once a week for 10 weeks with a circumference of 60 hours with mindfulness-based stress reduction and further process of the Mind / body medicine.
  Interventions: Behavioral: lifestyle-modification
- waiting control group (Active Comparator): A unique education unit within the scope of 3 hours on the influence of lifestyle factors on the disease and self-help materials for the independent training. After the follow-up measurement opportunity to participate in the program.
  Interventions: Behavioral: waiting control group

INTERVENTIONS:
Behavioral: lifestyle-modification — The group intervention is carried out once a week for 10 weeks for a total of 60 hours with elements of mindfulness-based stress reduction (MBSR) and further process of the mind / body medicine. In this project, this program will be adapted to the specific needs of crohn's disease patients.
  Arms: lifestyle-modification
Behavioral: waiting control group — Participants in this group receive a one-time education unit within the scope of 3 hours on the influence of lifestyle factors on the disease, also self-help materials for independent training offered. Following the follow-up measure also this group is given the opportunity to participate in the multimodal stress reduction- and lifestyle modification program.
  Arms: waiting control group

SUMMARY:
Patients with crohn's disease often suffer significant limitations to their quality of life, which are also conditioned by particular stress and psychosocial accompanying symptoms of the disease. A multimodal program for stress-reduction and lifestyle-modification has been shown to be effective in promoting the quality of life in patients with uncreative colitis. The study will examine the promotion of the quality of life of patients with crohn's disease and the positive Influence on stress, psychological symptoms and physiological parameters.

DETAILED DESCRIPTION:
40 patients with ulcerative colitis will be randomized in an Intervention group and a control group for 10 weeks. The primary outcome is the feasibility of the study, the intervention and the examinations. The Secondary outcomes are disease-specific quality of life, disease-activity, stress, psychological symptoms, inflammatory parameters, disease activity parameters, bowel parameter and the microbiome. As qualitative parameters, the influence of the disease on everyday life and the experience/ impact/ implementability of the programme will be investigated. Lastly, undesirable events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years
* Presence of a confirmed diagnosis of Crohn's disease
* In remission (not longer than 12 months, or mild to moderate clinical activity (HBI < 16)
* Medication that has been stable for at least 3 months, regardless of whether glucocorticoids, immunosuppressive drugs, azathioprine, or other drug treatments according to MBMCrohn - Version 1.0 from 06.12.2019 Page 7 Guideline
* Signed declaration of consent

Exclusion Criteria:

* infectious or refractory Crohn's disease with severe course
* Complete colectomy
* Severe psychological illness (e.g. depression requiring treatment, addiction, schizophrenia)
* Severe comorbid somatic disease (e.g. diabetes mellitus, oncological disease)
* Pregnancy
* Participation in stress reduction programmes or clinical studies on psychological interventions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Recruitment success | week 48
  Proportion of people responding to appeals for studies
Willingness to participate | week 48
  Proportion of people which actually agreed in relation to the proportion of people which responded to the appeal.
Attendance | week 48
  Proportion of people which actually attend the study
Loss of participants over the study period | week 48
  Proportion of people who quit during the study

SECONDARY OUTCOMES:
Disease-specific quality of life by IBD-Q | week 0
  Inflammatory Bowel Disease Questionnaire (IBD-Q), Recording on 7-point Likert scale, high values mean good, low values a reduced quality of life (1=worst score, 7=best score)
Disease-specific quality of life by IBD-Q | week 12
  Inflammatory Bowel Disease Questionnaire (IBD-Q), Recording on 7-point Likert scale, high values mean good, low values a reduced quality of life (1=worst score, 7=best score)
Disease-specific quality of life by IBD-Q | week 36
  Inflammatory Bowel Disease Questionnaire (IBD-Q), Recording on 7-point Likert scale, high values mean good, low values a reduced quality of life (1=worst score, 7=best score)
Disease-specific quality of life by IBD-Q | week 48
  Inflammatory Bowel Disease Questionnaire (IBD-Q), Recording on 7-point Likert scale, high values mean good, low values a reduced quality of life (1=worst score, 7=best score)
Generic quality of life by SF-36 | week 0
  Short Form Health 36 (SF-36) shows health-related quality of life, 36 items in 8 categories, 25% of the items must be filled in per category for evaluation. Lower sum score correlates with lower quality of life; higher sum score correlates with better quality of life.
Generic quality of life by SF 36 | week 12
  Short Form Health 36 (SF-36) shows health-related quality of life, 36 items in 8 categories, 25% of the items must be filled in per category for evaluation. Lower sum score correlates with lower quality of life; higher sum score correlates with better quality of life.
Generic quality of life by SF36 | week 36
  Short Form Health 36 (SF-36) shows health-related quality of life, 36 items in 8 categories, 25% of the items must be filled in per category for evaluation. Lower sum score correlates with lower quality of life; higher sum score correlates with better quality of life.
Generic quality of life by SF36 | week 48
  Short Form Health 36 (SF-36) shows health-related quality of life, 36 items in 8 categories, 25% of the items must be filled in per category for evaluation. Lower sum score correlates with lower quality of life; higher sum score correlates with better quality of life.
Disease activity 2 by BHI | week 0
  Harvey-Bradshaw Index - HBI is used to assess the degree of illness in individuals with Crohn's disease. The highest possible sum is 30 points and indicates a severe course of disease. A lower sum than 5 points indicates a clinical remission.
Disease activity by HBI | week 12
  Harvey-Bradshaw Index - HBI is used to assess the degree of illness in individuals with Crohn's disease. The highest possible sum is 30 points and indicates a severe course of disease. A lower sum than 5 points indicates a clinical remission.
Disease activity by HBI | week 36
  Harvey-Bradshaw Index - HBI is used to assess the degree of illness in individuals with Crohn's disease. The highest possible sum is 30 points and indicates a severe course of disease. A lower sum than 5 points indicates a clinical remission.
Disease activity by HBI | week 48
  Harvey-Bradshaw Index - HBI is used to assess the degree of illness in individuals with Crohn's disease. The highest possible sum is 30 points and indicates a severe course of disease. A lower sum than 5 points indicates a clinical remission.
Anxiety and depression by HADS | week 0
  Hospital Anxiety and Depression Scale (HADS), 14 items (7 each for depressive symptoms or symptoms of anxiety). The two summated scores of the summated scales HADS-A and HADS-D range between 0 and 21. high scores indicate depressivness and anxiety.
Anxiety and depression by HADS | week 12
  Hospital Anxiety and Depression Scale (HADS), 14 items (7 each for depressive symptoms or symptoms of anxiety). The two summated scores of the summated scales HADS-A and HADS-D range between 0 and 21. high scores indicate depressivness and anxiety.
Anxiety and depression by HADS | week 36
  Hospital Anxiety and Depression Scale (HADS), 14 items (7 each for depressive symptoms or symptoms of anxiety). The two summated scores of the summated scales HADS-A and HADS-D range between 0 and 21. high scores indicate depressivness and anxiety.
Anxiety and depression by HADS | week 48
  Hospital Anxiety and Depression Scale (HADS), 14 items (7 each for depressive symptoms or symptoms of anxiety). The two summated scores of the summated scales HADS-A and HADS-D range between 0 and 21. high scores indicate depressivness and anxiety.
Perceived stress by PSS | week 0
  Perceived Stress Scale (PSS), Rating on a five-step scale from 1 (=never) to 5 (=very often), high stress is assumed from a total score of 20 points
Perceived stress by PSS | week 12
  Perceived Stress Scale (PSS), Rating on a five-step scale from 1 (=never) to 5(=very often), high stress is assumed from a total score of 20 points
Perceived stress by PSS | week 36
  Perceived Stress Scale (PSS), Rating on a five-step scale from 1 (= never) to 5 (=very often), high stress is assumed from a total score of 20 points
Perceived stress by PSS | week 48
  Perceived Stress Scale (PSS), Rating on a five-step scale from 1 (= never) to 5 (=very often), high stress is assumed from a total score of 20 points
Coping strategies by COPE | week 0
  Coping Orientations to problems experienced Scale (COPE), total values of each scale vary between 2 (minimum) and 8 (maximum). Higher values indicate increased use of the specific coping strategy
Coping strategies by COPE | week 12
  Coping Orientations to problems experienced Scale (COPE), total values of each scale vary between 2 (minimum) and 8 (maximum). Higher values indicate increased use of the specific coping strategy
Coping strategies by COPE | week 36
  Coping Orientations to problems experienced Scale (COPE), total values of each scale vary between 2 (minimum) and 8 (maximum). Higher values indicate increased use of the specific coping strategy
Coping strategies by COPE | week 48
  Coping Orientations to problems experienced Scale (COPE), total values of each scale vary between 2 (minimum) and 8 (maximum). Higher values indicate increased use of the specific coping strategy
Flourishing by FS-D | week 0
  Flourishing Scale (FS-D), total value of the scale vary between 8 (minimum) and 56 (maximum). A high value corresponds to a person with many psychological resources and strengths.
Flourishing by FS-D | week 12
  Flourishing Scale (FS-D), total value of the scale vary between 8 (minimum) and 56 (maximum). A high value corresponds to a person with many psychological resources and strengths.
Flourishing by FS-D | week 36
  Flourishing Scale (FS-D), total value of the scale vary between 8 (minimum) and 56 (maximum). A high value corresponds to a person with many psychological resources and strengths.
Flourishing by FS-D | week 48
  Flourishing Scale (FS-D), total value of the scale vary between 8 (minimum) and 56 (maximum). A high value corresponds to a person with many psychological resources and strengths.
Core Self-Evaluation by CSES | week 0
  Core Self-Evaluation (CSES), 12 items on five-point Likert scale, 1 indicates disagreement and 5 indicates full agreement. High scores on the CSES represents a positive, confident, and self-efficacious person
Core Self-Evaluation by CSES | week 12
  Core Self-Evaluation (CSES), 12 items on five-point Likert scale, 1 indicates disagreement and 5 indicates full agreement. High scores on the CSES represents a positive, confident, and self-efficacious person
Core Self-Evaluation by CSES | week 36
  Core Self-Evaluation (CSES), 12 items on five-point Likert scale, 1 indicates disagreement and 5 indicates full agreement. High scores on the CSES represents a positive, confident, and self-efficacious person
Core Self-Evaluation by CSES | week 48
  Core Self-Evaluation (CSES), 12 items on five-point Likert scale, 1 indicates disagreement and 5 indicates full agreement. High scores on the CSES represents a positive, confident, and self-efficacious person
CRP (C-reactive protein) | week 0
  Determination of CRP in the blood
CRP (C-reactive protein) | week 12
  Determination of CRP in the blood
CRP (C-reactive protein) | week 36
  Determination of CRP in the blood
CRP (C-reactive protein) | week 48
  Determination of CRP in the blood
BSG (blood cell sedimentation rate) | week 0
  Determination of BSG in the blood
BSG (blood cell sedimentation rate) | week 12
  Determination of BSG in the blood
BSG (blood cell sedimentation rate) | week 36
  Determination of BSG in the blood
BSG (blood cell sedimentation rate) | week 48
  Determination of BSG in the blood
creatinin | week 0
  Determination of creatin in the blood
creatinin | week 12
  Determination of creatin in the blood
creatinin | week 36
  Determination of creatin in the blood
creatinin | week 48
  Determination of creatin in the blood
lymphocyte (T-cell) profiling | week 0
  Determination of lymphocyte (T-cell) profiling in the blood
lymphocyte (T-cell) profiling | week 12
  Determination of lymphocyte (T-cell) profiling in the blood
lymphocyte (T-cell) profiling | week 36
  Determination of lymphocyte (T-cell) profiling in the blood
calprotectin | week 0
  Determination of calprotectin in the stool
calprotectin | week 12
  Determination of calprotectin in the stool
calprotectin | week 36
  Determination of calprotectin in the stool
calprotectin | week 48
  Determination of calprotectin in the stool
lactoferrin | week 0
  Determination of lactoferrin in the stool
lactoferrin | week 12
  Determination of lactoferrin in the stool
lactoferrin | week 36
  Determination of lactoferrin in the stool
lactoferrin | week 48
  Determination of lactoferrin in the stool
(PMN)-elastase | week 0
  Determination of (PMN)-elastase in the stool
(PMN)-elastase | week 12
  Determination of (PMN)-elastase in the stool
(PMN)-elastase | week 36
  Determination of (PMN)-elastase in the stool
(PMN)-elastase | week 48
  Determination of (PMN)-elastase in the stool
Human beta-defensin-2 (hBD-2) | week 0
  Determination of hBD-2 in the stool
Human beta-defensin-2 (hBD-2) | week 12
  Determination of hBD-2 in the stool
Human beta-defensin-2 (hBD-2) | week 36
  Determination of hBD-2 in the stool
Human beta-defensin-2 (hBD-2) | week 48
  Determination of hBD-2 in the stool
zonulin | week 0
  Determination of zonulin in the stool
zonulin | week 12
  Determination of zonulin in the stool
zonulin | week 36
  Determination of zonulin in the stool
zonulin | week 48
  Determination of zonulin in the stool
alpha-1-antitrypsin | week 0
  Determination of alpha-antitrypsin in the stool
alpha-1- antitrypsin | week 12
  Determination of alpha-antitrypsin in the stool
alpha-1-antitrypsin | week 36
  Determination of alpha-antitrypsin in the stool
alpha-1-antitrypsin | week 48
  Determination of alpha-antitrypsin in the stool
intestinal microbiome | week 0
  Determination of intestinal microbiome
intestinal microbiome | week 36
  Determination of intestinal microbiome
Intestinal permeability | week 0
  confocal laser endomircoscopy
cortisol | week 12
  Determination of cortisol during Trier Social Stress Test at 4 points in time in the afternoon (right before, right after, 10 minutes after and 60 minutes after the Trier Social Stress Test)
ACTH | week 12
  Determination of ACTH during Trier Social Stress Test at 4 points in time in the afternoon (right before, right after, 10 minutes after and 60 minutes after the Trier Social Stress Test)
prolactin levels | week 12
  Determination of prolactin levels during Trier Social Stress Test at 4 points in time in the afternoon (right before, right after, 10 minutes after and 60 minutes after the Trier Social Stress Test)
glucocorticoid and β-adrenergic regulation of IL-8 and IL-10 | week 12
  Determination of glucocorticoid and β-adrenergic regulation of IL-8 and IL-10 during Trier Social Stress Test at 4 points in time in the afternoon (right before, right after, 10 minutes after and 60 minutes after the Trier Social Stress Test)
TNF-α production by peripheral blood cells | week 12
  Determination of TNF-α production by peripheral blood cells during Trier Social Stress Test at 4 points in time in the afternoon (right before, right after, 10 minutes after and 60 minutes after the Trier Social Stress Test)
heart rate | week 12
  Determination of heart rate during Trier Social Stress Test at 4 points in time in the afternoon (right before, right after, 10 minutes after and 60 minutes after the Trier Social Stress Test)
blood pressure systolic and diastolic | week 12
  Determination of blood pressure (systolic and diastolic) during Trier Social Stress Test at 4 points in time in the afternoon (right before, right after, 10 minutes after and 60 minutes after the Trier Social Stress Test)
STAI-S | week 12
  Determination of STAI-S during Trier Social Stress Test at 4 points in time in the afternoon (right before, right after, 10 minutes after and 60 minutes after the Trier Social Stress Test)
Adverse events | week 12
  all adverse events
Adverse events | week 36
  all adverse events
Adverse events | week 48
  all adverse events
qualitatives Interview | week 36
  guideline oriented qualitative interview about the influence of the disease on the patients' everyday life, experience with the programme offered, effects of the intervention on the disease, implementation of the intervention in everyday life
age (questionnaire) | week 0
  age in years
sex (questionnaire) | week 0
  identification of the gender (male/female)
weight | week 0
  weight in kilograms
body height | week 0
  body height in meters
School career (questionnaire) | week 0
  identification of the school career
job (questionnaire) | week 0
  identification of the actual job
professional career (questionnaire) | week 0
  identification of job qualifications
marital status (questionnaire) | week 0
  identification of the marital status (married/divorced/single/widowed)
occupation (questionnaire) | week 0
  identification of the type of occupation

CONTACTS AND LOCATIONS:
Overall Officials: Jost Langhorst, Prof., Study Director — Sozialstiftung Bamberg
Locations (1):
- Sozialstiftung Bamberg, Klinik für Intergrative Medizin, Bamberg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Schlee C, Uecker C, Oznur O, Bauer N, Langhorst J. Participants' perspectives on a multimodal stress management and comprehensive lifestyle modification program for patients with Crohn's disease-A qualitative interview study. PLoS One. 2024 Nov 13;19(11):e0313127. doi: 10.1371/journal.pone.0313127. eCollection 2024. PMID 39536026
- [Derived] Mekes-Adamczyk A, Gausmann N, Oznur O, Pfuhlmann K, Dziobaka J, Buer J, Langhorst J, Westendorf AM. Lifestyle Intervention Modulates the CD4+ T Cell Profile in the Blood of Crohn's Disease Patients. Inflamm Bowel Dis. 2025 Jan 6;31(1):200-209. doi: 10.1093/ibd/izae154. PMID 39102712
- [Derived] Bauer N, Loffler C, Oznur O, Uecker C, Keil T, Langhorst J. Mind-body-medicine and comprehensive lifestyle-modification in patients with Crohn's disease-Feasibility of a randomized controlled trial under pandemic circumstances. Front Integr Neurosci. 2022 Aug 23;16:960301. doi: 10.3389/fnint.2022.960301. eCollection 2022. PMID 36081609